CLINICAL TRIAL: NCT03797404
Title: Airway Remodeling Changes Induced by Mepolizumab in Severe Eosinophil Asthma
Brief Title: Airway Remodeling During Mepolizumab Treatment
Acronym: REMOMEPO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: GlaxoSmithKline (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: P180501J; 2018-002591-40 (EudraCT Number)
Record Dates: First submitted 2018-12-06; First posted 2019-01-09 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Asthma
Keywords: Eosinophil; Bronchial biopsies; Mepolizumab; Severe
MeSH Terms: conditions — Asthma; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mepolizumab: Patients receiving mepolizumab
- Patients w/o mepolizumab (retrospective): Retrospective control group of patients not exposed to mepolizumab, included in the COBRA cohort and the ASMATHERM protocol, who had 2 sets of biopsies and BAL within a 6 to 12 month-interval, without change in their treatment. Clinical data for this patients are available at inclusion and after 12 months.

SUMMARY:
Chronic airway changes, such as smooth muscle hypertrophy/hyperplasia, reticular basement membrane (RBM) thickening, goblet cells hyperplasia characterize severe asthma. Chronic inflammation, and especially eosinophilia and T2 cytokines are involved in these structural changes. The aim of this prospective observational study is to assess airway changes, assessed by bronchial biopsies before treatment, then after 6 months and 12 months, induced by mepolizumab in 40 severe asthma patients who will receive the treatment as part of their standard care. Changes in RBM thickening, in airway smooth muscle (ASM) area, in the number of PGP9 sections will be assessed on bronchial biopsies after 6 months and 12 months of mepolizumab treatment. Bronchoalveolar lavage (BAL) levels of inflammatory and remodeling mediators and of extra-cellular matrix (ECM) components will be measured after 6 months and 12 months of mepolizumab treatment. Relationship between clinical response to mepolizumab and remodeling changes after 6 months and 12 months will be assessed.

DETAILED DESCRIPTION:
1. Scientific Rationale & Hypothesis:

   Chronic airway changes, such as smooth muscle hypertrophy/hyperplasia, reticular basement membrane thickening, goblet cells hyperplasia characterize severe asthma. Chronic inflammation, and especially eosinophilia and T2 cytokines are involved in these structural changes. Increased ASM layer has been associated with eosinophilia for example, but not RBM thickening, suggesting that differential patterns of remodeling can be observed according to inflammatory patterns. Omalizumab, an anti IgE therapy, can reduce some features of airway remodeling, especially RBM and some parameters related to ASM. No data are available on potential changes in airway remodeling induced by mepolizumab.

   The aim of the study is to assess airway changes, assessed by bronchial biopsies, induced by mepolizumab in severe asthma patients who will receive the treatment as part of their standard care.

   All asthma patients refered to the asthma clinic are proposed to participate to the COBRA cohort (French national asthma cohort). Serum and DNA are collected at inclusion and every 6 months. Fiberoptic bronchoscopy (FOB) is routinely performed as part of the standard care for difficult-to-severe asthma in our centre for many years, to assess differential diagnosis and inflammatory pattern since Fractional exhaled nitric oxide (FeNO) is not routinely performed in France. BAL and 4 to 6 bronchial biopsies are performed.
2. Study Population:

   Severe asthma patients, refered to Severe Asthma Centre in Bichat and Bicetre Hospitals, receiving mepolizumab according to French recommendations (eos >300mm3 in the previous year, >2 exacerbations, despite optimal step 4-5 therapy, including daily use of steroids).
3. Study Design & Methods:

   * General study design Prospective, observational study in one Severe Asthma Centre : Bichat Hospital (Prof C.Taillé).

     40 patients will be prospectively included during a 32 months period.

This study aims to assess :

* Changes in RBM thickening, in ASM area after 6 months and 12 months of mepolizumab treatment
* Changes in BAL levels of inflammatory and remodeling mediators and of ECM components after 6 months and 12 months of mepolizumab treatment
* Changes in the number of PGP9 sections in the bronchial wall after 6 months and 12 months of mepolizumab treatment
* Relationship between clinical response to mepolizumab and remodeling changes after 6 months and 12 months of mepolizumab treatment
* Demographic and clinical characteristics of asthma (atopy, level of asthma control, FEV1…) will be available at inclusion and follow up, to assess clinical effect of mepolizumab treatment.

The following will perform at inclusion, 6 months and 12 months after initiating mepolizumab:

* clinical evaluation (age, BMI, atopic status, chronic rhinosinusitis, daily doses of steroids, exacerbations…)
* benefit of mepolizumab will be evaluated according to the physician's Global Evaluation of Treatment Effectiveness (GETE)
* asthma control test
* lung function test (FEV1, FEV1/VC, TLC, RV, pre/post salbutamol)
* FOB with BAL and 6 biopsies at inclusion, 6 months and 12 months
* Blood test for eosinophil count and serum conservation.

  * Study groups/arms Group 1 (prospective) : patients initiating a mepolizumab treatment. Group 2 (retrospective): to assess airway changes that can "spontaneously" occur during a 12 month-period, a retrospective "historical group" of patients included in the previous ASMATHERM study who had 2 sets of biopsies and BAL within a 6 to 12 month-interval, without exposure to mepolizumab and without change in their treatment during this interval, will be studied as a control group . Clinical data are available at inclusion and after 12 months.
  * Main tests or procedures All biopsies, BAL and serum analysis will be performed in the UMR1152 lab unit (Head: Dr Marina Pretolani).

Biopsies are fixed in formaldehyde and processed to paraffin wax for immunohistochemical (IHC) and morphometric studies. One biopsy will be stored at -80°C for further RNAseq analyses.

RBM thickening (morphometry), ASM area and the rate of ASM-proliferating cells (PCNA immuno-staining) will be measured. PGP9 staining can assess the number of nerves in the bronchial wall.

The number of inflammatory cells (eosinophils, neutrophils, mast cells, T-lymphocytes evaluated respectively by MBP, elastase, tryptase, CD4 expression) and vascular sections will also be enumerated after IHC. Eosinophils localization in the airway will be described.

Cytospin preparations from BAL cell pellets will be used to assess the proportion of eosinophils and neutrophils.

In parallel, the levels of different pro-inflammatory and remodeling mediators will be measured in BAL aliquots concentrated x 10, by specific Elisa and Luminex assays.

• Trial plan

V0: screening visit

V1: inclusion visit

* clinical evaluation
* Asthma control test
* Lung function test
* Fiber optic fibroscopy with BAL and bronchial biopsies (note that if a fiber optic fibroscopy with BAL and bronchial biopsies has already been performed in the month prior to inclusion, it will not be repeated at inclusion and the tissue and BAL samples will be retrieved for analysis)
* Blood sampling
* first treatment by Mepolizumab is administrated in the hospital.
* Patient injection training if this prescription is chosen
* Prescription for Mepolizumab, given at home for the next 6 months

V2: 6-month visit

* Clinical response assessment by GETE and ACT, clinical evaluation
* Lung function test
* Fiber optic fibroscopy with BAL and bronchial biopsies
* Blood sampling
* If responders, continuation of Mepolizumab treatment
* Compliance evaluation (file signed by the nurse or patient after each injection)

V3: 12-month visit

* clinical response assessment by GETE and ACT, clinical evaluation
* Lung function test
* Fiber optic fibroscopy with BAL and bronchial biopsies
* Blood sampling
* Compliance evaluation (file signed by the nurse or patient after each injection)

ELIGIBILITY:
Inclusion criteria:

* adult >18 years,
* severe uncontrolled asthma, defined as eosinophil blood count >300/mm3 in the previous 12 months and at least 2 exacerbations in the previous 12 months or requiring oral steroids for more than half of the previous year,
* indication for mepolizumab decided by an asthma specialist,
* efficient contraception, for women of reproductive age

Exclusion criteria :

* pregnancy,
* smokers or ex smokers >10 pack/yr,
* contra indication for fiberoptic bronchoscopy (allergy to xylocain, antiaggregant or anticoagulant treatment...),
* contra indication for mepolizumab,
* patient who previously received mepolizumab or already received mepolizumab at inclusion,
* participation in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe uncontrolled eosinophil asthma with an indication for mepolizumab according to French recommandations (eos >300mm3 in the previous year, >2 exacerbations, despite optimal step 4-5 therapy, including daily use of steroids).
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Changes in reticular basement membrane (RBM) thickening | 0, 6 and 12 months
  The absolute variation in RBM thickening (µm, morphometry measurement on bronchial biopsies) over 12 months is defined as the difference between month twelve and baseline (V1).
  The absolute variation in RBM thickening over 6 months is defined as the difference between month six and baseline (V1).
Changes in airway smooth muscle (ASM) area | 0, 6 and 12 months
  Measured in morphometry in µm2 and expressed as a percentage of smooth muscle surface area relative to the biopsy surface.
  The absolute variation in ASM area over 12 months is defined as the difference between month twelve and baseline (V1).
  The absolute variation in ASM area over 6 months is defined as the difference between month six and baseline (V1).
Number of proliferating muscle cells | 0, 6 and 12 months
  Evaluated by anti proliferating cell nuclear antigen (PCNA) antibodies, expressed as the number of positive cells per muscle surface.
Number of nerve endings | 0, 6 and 12 months
  Evaluated by PGP9 and expressed as number of positive cells per biopsy surface in mm2
Number of vascular sections | 0, 6 and 12 months
  Measured with an anti-CD31 antibody, expressed in number of sections per mm2.
Number of infiltrating inflammatory cells in the biopsies | 0, 6 and 12 months
  Number of infiltrating inflammatory cells (infiltrating neutrophils, lymphocytes and eosinophils) expressed as number of positive cells per biopsy surface in mm2
Number of inflammatory cells in the BAL | 0, 6 and 12 months
  Number of inflammatory cells (neutrophils, lymphocytes and eosinophils) expressed as % of total cells in the BAL
Proportion of eosinophils expressing MBP/IL3R | 0, 6 and 12 months
  Measured on bronchial biopsies, expressed as number of cells per biopsy surface in mm2

SECONDARY OUTCOMES:
Interferon-gamma concentration | 0, 6 and 12 months
  Interferon-gamma (Th1 cytokine) will be measured in BAL and serum
IL-13 concentration | 0, 6 and 12 months
  IL-13 (Th2 cytokine) will be measured in BAL and serum
Periostin concentration | 0, 6 and 12 months
  Periostin (Th2 cytokine) will be measured in BAL and serum
IL-17A concentration | 0, 6 and 12 months
  IL-17A (Th17 cytokine) will be measured in BAL and serum
IL-22 concentration | 0, 6 and 12 months
  IL-22 (Th17 cytokine) will be measured in BAL and serum
IL-33 concentration | 0, 6 and 12 months
  IL-33 (innate immune cytokines) will be measured in BAL and serum
Thymic Stromal Lymphopoietin (TSLP) concentration | 0, 6 and 12 months
  TSLP (innate immune cytokines) will be measured in BAL and serum
Fibronectin concentration | 0, 6 and 12 months
  Fibronectin (soluble hallmarks of ECM remodeling) will be measured in BAL and serum
Tenascin concentration | 0, 6 and 12 months
  Tenascin (soluble hallmarks of ECM remodeling) will be measured in BAL and serum
Fibulin-1 concentration | 0, 6 and 12 months
  Fibulin-1 (soluble hallmarks of ECM remodeling) will be measured in BAL and serum
Monocyte chemoattractant protein-1 (CCL/MCP-1) concentration | 0, 6 and 12 months
  Will be measured in BAL and serum
EGF concentration | 0, 6 and 12 months
  Will be measured in BAL and serum
bFGF concentration | 0, 6 and 12 months
  Will be measured in BAL and serum
PDGF-BB concentration | 0, 6 and 12 months
  Will be measured in BAL and serum
Total score at Asthma Control Test | 0, 6 and 12 months
  Measured using the Asthma Control Test (ACT) scale (range: 5 to 25). ACT assesses the frequency of shortness of breath and general asthma symptoms, use of rescue medications, the effect of asthma on daily functioning, and overall self-assessment of asthma control.
  * 5 items, with 4-week recall (on symptoms and daily functioning)
  * each item is evaluated by a 5-point scale (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled).
  The total score ranges from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.
Global evaluation of mepolizumab benefit | 6 and 12 months
  Benefit of mepolizumab will be evaluated by patient and by physician according to the physician's Global Evaluation of Treatment Effectiveness (GETE).
  Patients will be considered as "responders" if classified as "excellent response" or "good response" by their physician.
Forced expiratory volume (FEV1) | 0, 6 and 12 months
  Measured during lung function test, pre/post salbutamol, expressed in ml.
Forced expiratory volume (FEV1) | 0, 6 and 12 months
  Measured during lung function test, pre/post salbutamol, expressed in % of predicted value.
Forced expiratory volume/Vital capacity (FEV1/VC) | 0, 6 and 12 months
  Measured during lung function test, pre/post salbutamol, expressed in %
Total lung capacity (TLC) | 0, 6 and 12 months
  Measured during lung function test, pre/post salbutamol, expressed in ml.
Total lung capacity (TLC) | 0, 6 and 12 months
  Measured during lung function test, pre/post salbutamol, expressed in % of predicted value.
Residual volume (RV) | 0, 6 and 12 months
  Measured during lung function test, pre/post salbutamol, expressed in ml.
Residual volume (RV) | 0, 6 and 12 months
  Measured during lung function test, pre/post salbutamol, expressed in % of predicted value.
Proportion of patients with pre-bronchodilator FEV1 greater than 80% | 6 and 12 months
  In order to assess functional response to treatment
Proportion of patients with an increase from baseline in pre-bronchodilator FEV1 greater than 20% | 6 and 12 months
  In order to assess functional response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Camille TAILLE, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Bichat hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Taille C, Hamidi F, Heddebaut N, Pote N, Le Guen P, Le Brun M, Roy C, Dupont A, Letuve S. Impact of Mepolizumab on Airway Remodeling and Inflammation in Severe Eosinophilic Asthma. Chest. 2025 Dec 5:S0012-3692(25)05814-3. doi: 10.1016/j.chest.2025.10.047. Online ahead of print. PMID 41354402